CLINICAL TRIAL: NCT00907218
Title: An Open Pilot Study of Varenicline (Chantix) in Adult Smokers With Attention Deficit Hyperactivity Disorder (ADHD): Effects on ADHD and Cigarette Smoking
Brief Title: Chantix in Adult Smokers With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: extremely slow enrollment
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Timothy Wilens, MD, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-P-000444
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Results first posted 2013-09-23 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-09

CONDITIONS: Attention Deficit/Hyperactivity Disorder; Smoking Cessation
Keywords: ADHD; Attention Deficit Hyperactivity Disorder; ADHD medication; Chantix; varenicline; smoking; smoking cessation; quit smoking
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Smoking Cessation; Smoking | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Adults who meet DSM-IV-TR criteria for ADHD and smoke cigarettes.
  Interventions: Drug: Varenicline (Chantix)

INTERVENTIONS:
Drug: Varenicline (Chantix) — Upon completion of screening procedures and meeting eligibility criteria, subjects will begin taking varenicline daily until Week 6 of the study. At Week 6 they will discontinue varenicline and return one week later for their final study visit to assess return of ADHD symptomatology. Subjects will start on 0.5 mg of varenicline per day for the first week of treatment. The dose will be increased to 0.5 mg twice a day at the end of week 1 visit, and then increased to 1 mg twice a day at the end of week 2 visit, to remain at this dose until the week 6 visit. At week 6, all subjects will be openly discontinued from varenicline, to return to the office the following week for re-assessment one week off the medication. If significant adverse effects (AE) occur, the daily dose may be reduced by 0.5 to 1 mg. At subsequent visits, a higher dose may be resumed if tolerated. Maximum dose will be 2 mg daily.
  Other Names: Chantix(varenicline) is a smoking cessation medicine.

SUMMARY:
The purpose of this research study is to learn about the efficacy of a medication called varenicline (Chantix) in treating ADHD in adults and in reducing cigarette smoking in adults with ADHD. The investigators hypothesize that ADHD symptomatology in adults with ADHD will be improved with varenicline treatment. The investigators also hypothesize that varenicline treatment will result in significant reductions in cigarette smoking. Another objective of this study is to more fully evaluate the response and tolerability to varenicline in this group of cigarette smoking adults with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients from 18-60 years of age;
* A cigarette smoking history of at least 3 months, and currently smoking;
* An interest in quitting smoking and a willingness to comply with all study procedures and medication instructions;
* A current DSM-IV-TR diagnosis of ADHD confirmed by clinical psychiatric evaluation and/or ADHD module of structured diagnostic interview, completed by study clinician.
* For females of child-bearing potential: pregnancy test at screening visit is negative and the subject does not plan to become pregnant during the study.

Exclusion Criteria:

* Pregnancy or breast-feeding;
* Clinically significant and/or unstable medical condition including renal, hepatic, or neurological, based upon a medical history and vital signs;
* Ongoing treatment with medications which may be affected (altered blood levels) if subjects stop smoking in the study, including insulin, theophylline, and blood thinners, as determined by clinician;
* Clinically significant cardiovascular history, including myocardial infarction, untreated hypertension, atrial fibrillation, or arrhythmia;
* Current untreated psychiatric comorbidity which the investigator judges to be of greater than mild severity, including Major Depressive Disorder;
* Current psychiatric comorbidity, including suicidality, homicidality, psychosis, determined by the clinician to be clinically significant and/or unstable
* Lifetime history of DSM-IV Bipolar I disorder, Schizophrenia, or suicide attempt as determined through clinical evaluation or diagnostic interview;
* Currently (within 3 months) meets DSM-IV criteria for abuse or dependence for any psychoactive substance other than nicotine;
* Current treatment with mood stabilizers, anti-psychotics, nicotine replacement therapies, or varenicline;
* Mental retardation (IQ < 75);
* History of intolerance or allergy to varenicline.
* Clinically significant abnormal screening values including:

  * Consistent readings of hypertension (>140/90) during screening period (including screening and baseline visits), defined as two or more readings (each being the average of three measurements) at a single visit with systolic blood pressure, SBP > 140 and/or diastolic blood pressure, DBP, > 90, and confirmed by manual reading.

Subjects with isolated incidences (of triplicate average BP) of SBP > 140 and/or DBP > 90 at baseline/week 0 visit, confirmed by manual reading, which are determined to be clinically significant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Wilens, MD, Principal Investigator — Massachusetts General Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 studies were recruited. They participated in a previous study in our department and signed consent for the data to be used for this study.
Pre-assignment Details: Recruitment was extremely slow and therefore the study was terminated early
Groups:
- Adults Who Meet DSM-IV-TR Criteria for Attention Deficit Hyper: Varenicline (Chantix) : Upon completion of screening procedures and meeting eligibility criteria, subjects will begin taking varenicline daily until Week 6 of the study. At Week 6 they will discontinue varenicline and return one week later for their final study visit to assess return of ADHD symptomatology. Subjects will start on 0.5 mg of varenicline per day for the first week of treatment. The dose will be increased to 0.5 mg twice a day at the end of week 1 visit, and then increased to 1 mg twice a day at the end of week 2 visit, to remain at this dose until the week 6 visit. At week 6, all subjects will be openly discontinued from varenicline, to return to the office the following week for re-assessment one week off the medication. If significant adverse effects (AE) occur, the daily dose may be reduced by 0.5 to 1 mg. At subsequent visits, a higher dose may be resumed if
Period: Overall Study
Arm/Group | Adults Who Meet DSM-IV-TR Criteria for Attention Deficit Hyper
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | No Data Was Analyzed
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: The DSM-IV Based Adult ADHD Investigator Symptom Rating Scale (AISRS)
Description: The AISRS is an 18-item questionnaire administered by the clinician assessing each of the individual DSM-IV symptoms of ADHD. Each symptom is rated on a scale of severity from 0 (none) to 3 (severe), and the 18 symptom questions are summed to calculate a total score. The minimum total score is a 0, while the maximum total score is a 54.
Time Frame: Weekly for 7 weeks
Population: Data was not collected due to study termination, 2 subjects were recruited however their data was not analyzed
Groups:
- Adults Who Meet DSM-IV-TR Criteria for ADHD and Smoke Cigarett: Varenicline (Chantix): Upon completion of screening procedures and meeting eligibility criteria, subjects will begin taking varenicline daily until Week 6 of the study. At Week 6 they will discontinue varenicline and return one week later for their final study visit to assess return of ADHD symptomatology. Subjects will start on 0.5 mg of varenicline per day for the first week of treatment. The dose will be increased to 0.5 mg twice a day at the end of week 1 visit, and then increased to 1 mg twice a day at the end of week 2 visit, to remain at this dose until the week 6 visit. At week 6, all subjects will be openly discontinued from varenicline, to return to the office the following week for re-assessment one week off the medication. If significant adverse effects (AE) occur, the daily dose may be reduced by 0.5 to 1 mg. At subsequent visits, a higher dose may be resumed if tolerated. Maximum dose will be 2 mg daily.
Arm/Group | Adults Who Meet DSM-IV-TR Criteria for ADHD and Smoke Cigarett
Number analyzed (Participants) | 0

2. Primary Outcome: Time Line Follow Back of Cigarette Smoking
Description: The reduction in cigarette smoking, defined as the change from baseline on the amount of cigarettes per day smoked (cpd), using the time-line follow back method. This method involves asking subjects to retrospectively estimate their cigarette use 7 days to 2 years prior to the interview date.
Time Frame: Weekly for 7 weeks
Population: Data was not collected due to study termination, 2 subjects were recruited however their data was not analyzed
Arm/Group | Adults Who Meet DSM-IV-TR Criteria for ADHD and Smoke Cigarett
Number analyzed (Participants) | 0

3. Secondary Outcome: Exhaled CO Levels
Description: At baseline and all weekly study visits,exhaled carbon monoxide (CO) levels were read.
Time Frame: Weekly over 7 weeks
Population: Data was not collected due to study termination, 2 subjects were recruited however their data was not analyzed
Arm/Group | Adults Who Meet DSM-IV-TR Criteria for ADHD and Smoke Cigarett
Number analyzed (Participants) | 0

4. Secondary Outcome: Rates of Smoking Cessation
Description: Varenicline has efficacy in smoking sensation; therefore smoking cessation was measured at baseline and at all study visits.
Time Frame: Weekly for 7 weeks
Population: Data was not collected due to study termination, 2 subjects were recruited however their data was not analyzed
Arm/Group | Adults Who Meet DSM-IV-TR Criteria for ADHD and Smoke Cigarett
Number analyzed (Participants) | 0

5. Secondary Outcome: ADHD Clinical Global Impressions Scale Improvement (CGI-I) and Severity (CGI-S)
Description: The Clinical Global Impression Scale of ADHD for Improvement and Severity assess overall severity and change in severity of ADHD. The CGI-I scale is rated from 1 to 7 (1=very much improved; 7=very much worse). The CGI-S is rated from 1 to 7 as well (1=not ill; 7=extremely ill).
Time Frame: Weekly for 7 weeks
Population: Data was not collected due to study termination, 2 subjects were recruited however their data was not analyzed
Arm/Group | Adults Who Meet DSM-IV-TR Criteria for ADHD and Smoke Cigarett
Number analyzed (Participants) | 0

6. Secondary Outcome: Vital Signs
Description: Vital signs were collected at each study visit, including height, weight, blood pressure, and heart rate.
Time Frame: Weekly for 7 weeks
Population: Data was not collected due to study termination, 2 subjects were recruited however their data was not analyzed
Arm/Group | Adults Who Meet DSM-IV-TR Criteria for ADHD and Smoke Cigarett
Number analyzed (Participants) | 0

7. Secondary Outcome: Spontaneous Reports of Adverse Effects
Description: Reports of adverse events were completed at baseline and weekly visits throughout the trial.
Time Frame: Weekly for 7 weeks
Population: Data was not collected due to study termination, 2 subjects were recruited however their data was not analyzed
Arm/Group | Adults Who Meet DSM-IV-TR Criteria for ADHD and Smoke Cigarett
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: adverse event data was not collected
Description: only 2 subjects were recruited and they had previously participated in a study and we used the data for that study. Therefore there was no adverse events
Arm/Group | Adults Who Meet DSM-IV-TR Criteria for Attention Deficit Hyper
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Extremely slow enrollment so the study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No